CLINICAL TRIAL: NCT01922531
Title: Defining Axonal Injury in Children With Mild Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CCHMC001
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Traumatic Brain Injury
Keywords: mTBI; Mild Traumatic Brain Injury; Axonal Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mild Traumatic Brain Injury: These were patients who presented to the ER within 6 hours of a witnessed head injury. Patients were also eligible if the patient had a self-reported head injury with evidence of head trauma.
- Orthopedic Injury: Patients were eligible as an orthopedic injured control who presented to the ER within 6 hours of an isolated extremity trauma that radiography and an Abbreviated Injury Scale (AIS) of less than or equal to 3.

SUMMARY:
To measure Axonal Injury in children with mild traumatic brain injury enrolled in an Emergency Department using Diffusion Tensor Imaging, a type of MRI and biomarkers.

DETAILED DESCRIPTION:
Objective: To determine if children with mild traumatic brain injury (mTBI) have acute axonal injury defined by disruption of diffusion of water in white matter using diffusion tensor imaging (DTI) as compared to orthopedic injury (OI) controls.

Methods: Children ages 11-16 years who presented within 6 hours of either a mTBI or an isolated OI were recruited from the emergency department (ED). Patients had Diffusion Tensor Imaging (DTI) study performed within 96 hours of injury. Voxel based analysis approach was used to quantify the group differences for common DTI measures. In the ED and at the time of the scan, symptom burden was measured using the post concussion symptom scale.

ELIGIBILITY:
Inclusion Criteria:

mTBI group: Inclusion: Children between the ages of >11 to < 16 years who present within 6 hours of injury with a witnessed head injury. A patient may have a self-reported injury to the head but there must also be evidence of head trauma on exam to be eligible for the study. Subjects must meet the clinical definition of mTBI from the American Congress of Rehabilitation Medicine122: A blow to the head or acceleration/deceleration movement of the head resulting in one or more of the following: i. loss of consciousness <30 minutes, ii. amnesia <24 hours, iii. any alteration in mental state at the time of the injury. Subjects without witnessed LOC/amnesia but with demonstrable amnesia in the ED are eligible. Subject must have GCS of 13-15 at the time of arrival in the ED. Subject may be enrolled prior to CT (if completed). Subjects should only have up to 1 other minor extracranial injury defined by an Abbreviated Injury Severity Scale < 1 to that region (AIS; American Association for Automotive Medicine, 1990). Subjects will be included if they have multiple injuries that affect only 1 body system as noted in the AIS (ie, subjects who sustain skin abrasions to more than 1 body region as a result of injury but do not meet exclusion based on injury severity) Subjects and their families must be able to speak and read English. Subjects must agree to have blood drawn in the ED, and to return three times as an outpatient for repeat testing. Subjects are still eligible if they are admitted to the hospital. Subjects must have a score of less than 65 on the CBCL to be included in the study to limit possible co-morbidities. Children with a diagnosis of Attention Deficit / Hyperactivity Disorder (ADHD) will be included as long as they meet the following criteria: physician diagnosed, controlled by only one ADHD medication, and have a T-score of less than 50 on the DSM Oriented Scale for Attention Deficit / Hyperactivity Disorder (Sub-Category of CBCL).

Orthopedic Injury Control Group:

Subjects with isolated extremity trauma requiring radiography and an Abbreviated Injury Scale (AIS) of < 3 (AIS; American Association for Automotive Medicine, 1990)123 will be included in the study. The presence of a fracture on the x-ray is not a requirement for inclusion. Subjects can not require immediate surgery for care. We will attempt to match based on gender and age (+/- 365 days within the included age range 11-16); yet, we will enroll consecutive eligible patients meeting inclusion/exclusion criteria.Subjects must not have any evidence of head trauma / facial trauma or symptoms of concussion (such as LOC, amnesia, confusion). This information must be corroborated with a reliable witness or the parent and the treating physician. Subjects must have normal neurologic exams and must not require a head CT as a part of the clinical care. Subjects may be prescribed narcotics and/or opiates prescribed for pain in the ED will be allowed IF the subject agrees to refrain from taking the medication for at least 4 hours prior to completing the neurobehavioral testing at follow-up. Subjects must meet the same CBCL score and ADHD definition as listed in the mTBI group.

Exclusion Criteria:

mTBI Group: Exclusion Criteria: Children <11 or >16 years old and subjects and/or the families do not speak and read English will be excluded. Subjects with a score of 65 or more on the CBCL will be excluded due to probable pre-existing impairment. Any subject who has an altered mental status due to the ingestion of substances of abuse or alcohol or who are prescribed a drug that impairs cognition (e.g., benzodiazepines, antipsychotics, or opiates such as those listed (but not limited to) in Appendix L). Subjects will be excluded if they have a prior history of concussion, pre-existing neurologic impairment (stroke, prior TBI requiring ED visit or hospitalization, CSF shunt, brain tumor), pre-existing cognitive disorders (seizure disorder, mental retardation), psychological problems or developmental delay. Subjects with the following illnesses will also be excluded: bleeding or coagulation disorders, cancer (who are currently undergoing treatment), HIV/AIDS, schizophrenia, multiple sclerosis, cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy (CADASIL), amyotrophic lateral sclerosis (ALS), Alzheimer's Disease, Creutzfeldt-Jakob Disease, and Krabbe Disease. Subjects will be excluded if they have the diagnosis of ADHD and require 2 or more medications for control or they have a T-score of 50 or greater on the DSM Oriented Scale for Attention Deficit / Hyperactivity Disorder. Subjects will be excluded if they are on any medication typically prescribed for ADHD but do not carry the diagnosis of ADHD. Subjects will be excluded if they have any condition that precluded them from undergoing magnetic resonance imaging as detailed in Appendix L. These include having an implanted medical devices (i.e., cardiac pace maker, hearing aid, or other implant); having metal in the body that does not meet criteria for MRI machines (i.e. braces, plates, screws; since some types of metal are not responsive to the magnet and are permitted, the eligibility for MRI will be investigated in each such case to ensure safety); having non-removable jewelry or body piercing; pregnancy; known claustrophobia; extreme obesity (due to physical limitation of the magnet). Subjects with one extracranial (organ group) injury with an AIS score of > 2 or 2 or more extracranial (i.e. 2 or more organ groups) injuries will be excluded, those with multiple injuries to one organ group (ie, skin abrasion on more than 1 extremity) will still be eligible.

Orthopedic Injury Control Group:

Subjects who present with an orthopedic injury, as well as head trauma or signs or symptoms of mTBI will be excluded. Subjects who do not have a reliable witness to determine that there was no loss of consciousness, amnesia, or confusion related to the injury will be excluded. Subjects who are enrolled then subsequently receive a Head CT will have enrollment discontinued. Subjects who are prescribed a drug that impairs cognition (e.g., benzodiazepines, antipsychotics, opiates) will be excluded. Any inability or unwillingness to complete study procedures including follow up procedures will be excluded. Subjects will not be eligible to serve as controls if they cannot use a computer mouse due to their injury. Patients must not have any of the other exclusion criteria listed for the mTBI group (ie, CBCL scores, ADHD diagnosis, pre-existing conditions,MRI Contraindications)

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients presenting to a Pediatric Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Differences in mean FA | 72 hours post enrollment
  The primary analysis was to test for significant differences in mean Fractional Anisotropy in the Corpus Callosum between the mild traumatic brain injured patients and orthopedic controls.

SECONDARY OUTCOMES:
Functional Outcomes following mTBI | 1 week and 1 month post injury
  Four meausres were used to assess functional outcomes following mTBI. These were completed at 1 week and 1 month post injury.

OTHER OUTCOMES:
Biomarkers | 6 hours post injury
  Participants with mTBI and OI had blood drawn up to 6 hours post injury to analyze the differences in serum proteomes to identify known and novel biomarkers of axonal injury associated with mild traumatic brain injury in children.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Babcock, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States